CLINICAL TRIAL: NCT01438177
Title: A Phase II, Trial of Chloroquine in Combination With VELCADE and Cyclophosphamide in Patients With Relapsed and Refractory Myeloma
Brief Title: Chloroquine in Combination With VELCADE and Cyclophosphamide for Relapsed and Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution.
Sponsor: NYU Langone Health (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-02008
Record Dates: First submitted 2011-09-08; First posted 2011-09-21 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Multiple Myeloma
Keywords: myeloma; multiple myeloma; relapsed myeloma; refractory myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Bendamustine Hydrochloride; Cyclophosphamide; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Velcade+Cyclophosphamide+Chloroquine (Experimental): VELCADE given by intravenous push at 1.3 mg/m^2 on days 1, 4, 8, 11, 22, 25, 29 and 32.
  Cyclophosphamide given at 50 mg orally twice per day on days 1-14 and 22-35.
  Chloroquine given at 500 mg orally daily on days 1-14 and 22-35.
  Each cycle is 42 days in length.
  Interventions: Drug: Velcade; Drug: Cyclophosphamide; Drug: Chloroquine

INTERVENTIONS:
Drug: Velcade
  Other Names: Bendamustine HCl; Treanda; Bortezomib
Drug: Cyclophosphamide
  Other Names: Cytoxan; Neosar; Endoxan; Revimmune; Procytox
Drug: Chloroquine
  Other Names: Aralen

SUMMARY:
This pilot phase II trial studies how well giving bortezomib and cyclophosphamide together with chloroquine works in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Chloroquine may help chemotherapy drugs work better by making cancer cells more sensitive to the drug. Giving bortezomib and cyclophosphamide together with chloroquine may kill more cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. Female subject is either post-menopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of VELCADE, or agree to completely abstain from heterosexual intercourse. Male subjects, even if surgically sterilized (ie, status postvasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.
3. Diagnosis of multiple myeloma based on standard criteria as follows:

   Major Criteria:

   I. Plasmacytomas on tissue biopsy

   II. Bone marrow plasmacytosis (>30% plasma cells)

   III. Monoclonal immunoglobulin spike on serum electrophoresis (IgG >3.5 G/dL or IgA > 2.0 G/dL) or kappa or lambda light chain excretion> 1 G/day on 24 hour urine protein electrophoresis

   Minor Criteria
   1. Bone marrow plasmacytosis (10 to 30% plasma cells)
   2. Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria
   3. Lytic bone lesions
   4. Normal IgM < 50 mg/dL, IgA < 100 mg/dL, or IgG < 600 mg/dL

   Any of the following sets of criteria will confirm the diagnosis of Multiple Myeloma:
   * Any two of the major criteria
   * Major criterion I plus minor criterion b, c, or d
   * Major criterion III plus minor criterion a or c
   * Minor criteria a, b and c or a, b and d
4. Measurable disease, defined as a monoclonal immunoglobulin spike on serum electrophoresis of ≥ 1 Gm/dL and/or urine monoclonal immunoglobulin spike of ≥ 200 mg/24 hours.
5. Patients must have refractory myeloma as defined by a greater than 25% increase in their M-protein. They should have progressed on a combination of VELCADE and cyclophosphamide.
6. Non-secretors must have measurable protein by Freelite or measurable disease such as plasmacytoma to be eligible.
7. Karnofsky performance status ≥ 50
8. Patients treated with local radiotherapy with or without a brief exposure to steroids are eligible. Patients who require concurrent radiotherapy should have entry to the protocol deferred until the radiotherapy is completed
9. Meets the following pretreatment laboratory criteria at Baseline (Day 1 of Cycle 1, before study drug administration)

   * Absolute neutrophil count ≥ 0.5 x 10^3/uL
   * Calculated or measured creatinine clearance ≥ 30 mL/min
10. Age 18 years or older

Exclusion Criteria:

1. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes)
2. Plasma cell leukemia
3. Receiving steroids daily for other medical conditions, e.g., asthma, systemic lupus erythematosis, rheumatoid arthritis
4. Infection not controlled by antibiotics
5. HIV infection. Patients should provide consent for HIV testing according to the institution's standard practice
6. Known active hepatitis B or C
7. Patient had myocardial infarction within 6 months prior to enrollment, New York Hospital Association (NYHA) Class III or IV heart failure, (see appendix D), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
8. Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
9. Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.
10. Other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol
11. Female subject is pregnant or lactating. Confirmation that the subject is not pregnant must be established by a negative serum B-human chorionic gonadotropin (B hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for postmenopausal or surgically sterilized women.
12. Patient has > Grade 2 peripheral neuropathy
13. Patient has known hypersensitivity to VELCADE, boron or mannitol, quinidine or quinidine derivatives or to cyclophosphamide or any component of the formulation.
14. Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
15. Patients with preexisting retinal or visual field changes.
16. Patient has > 1.5 x upper limit of normal Total Bilirubin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grossbard, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Cancer Institute, New York, New York, United States

REFERENCES:
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From Oct. 2011 to March 2013, 11 patients were enrolled to the study from New York University Langone Medical Center.
Period: Overall Study
Arm/Group | Velcade+Cyclophosphamide+Chloroquine
Started | 11
Completed | 9 (Patients who were off due to disease progression)
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Initiation of new therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Velcade+Cyclophosphamide+Chloroquine
Number analyzed (Participants) | 11
Age, Customized [Number; unit: participants]
  45-53 years | 2
  54-63 years | 4
  64-73 years | 4
  74-83 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (CR + PR After 2 Cycles)
Description: Response rate is defined as the percentage of patients who have a complete response (CR) or partial response (PR). Responses were assessed every two cycles of treatment, based on the criteria published by the International Myeloma Working Group (Durie, et al, 2006). Per International Myeloma Working Group response criteria:
  CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow PR: > 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or to < 200 mg/24 h
Time Frame: Up to 2 years
Population: Evaluable patients.
Measure: Number; unit: percentage of participants
Arm/Group | Velcade+Cyclophosphamide+Chloroquine
Number analyzed (Participants) | 9
percentage of participants | 30

2. Secondary Outcome: Number of Participants With Adverse Events of Grade 3 or Higher
Description: Adverse events reported here were at least possibly related to the protocol therapy.
Time Frame: Treatment period plus 30 days post-treatment
Population: Any patients who started the treatment
Measure: Number; unit: participants
Arm/Group | Velcade+Cyclophosphamide+Chloroquine
Number analyzed (Participants) | 9
participants
  Fatigue | 2
  Hemoglobin | 1
  Nasal cavity/paranasal reactions | 1
  ANC/AGC | 4
  Pain: pleural | 1
  Platelets | 5

3. Secondary Outcome: Percentage of Subjects Who Have Complete Response or Partial Response and Have 2+ or Higher Autophagy
Time Frame: until clinical response (up to 2 years)
Population: Study was terminated prior to collection of this data point.
Arm/Group | Velcade+Cyclophosphamide+Chloroquine
Number analyzed (Participants) | 0

4. Secondary Outcome: Median Duration of Response of This Regimen
Description: Duration of response is the time from response (CR or PR) until progression of disease or relapse. Responses and progression were evaluated based on the criteria published by the International Myeloma Working Group (Durie, et al, 2006).
Time Frame: up to 2 years
Population: patients who have responded
Measure: Median (Full Range); unit: months
Arm/Group | Velcade+Cyclophosphamide+Chloroquine
Number analyzed (Participants) | 9
months | 4.4 [3.9 to 8.3]

ADVERSE EVENTS:
Time Frame: During treatment and within 30 days post-treatment
Description: All adverse events were reported regardless of attribution to protocol therapy.
Arm/Group | Velcade+Cyclophosphamide+Chloroquine
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade+Cyclophosphamide+Chloroquine (N=11)
pain: pleura (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade+Cyclophosphamide+Chloroquine (N=11)
Anorexia (Gastrointestinal disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 1
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Creatinine (Investigations) | 1
Dehydration (Gastrointestinal disorders) | 1
Dental: teeth (Gastrointestinal disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Distension/bloating, abdominal (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 2
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Edema: limb (Blood and lymphatic system disorders) | 1
Eyelid dysfunction (Eye disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 10
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L): (General disorders) | 1
Flu-like syndrome (Infections and infestations) | 3
Fracture (Musculoskeletal and connective tissue disorders) | 2
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 2
Infection - Other: ocular Hepes (Infections and infestations) | 1
Infection - Other: shingles (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Eye NOS (Infections and infestations) | 1
Infection with unknown ANC: Skin (cellulites) (Infections and infestations) | 1
Insomnia (General disorders) | 2
Metabolic/Laboratory - Other: high BUN (Investigations) | 1
Mood alteration: Agitation (Nervous system disorders) | 1
Mood alteration: Depression (Nervous system disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 4
Nausea (Gastrointestinal disorders) | 7
Neuropathy: sensory (Nervous system disorders) | 5
Neutrophils/granulocytes (ANC/AGC): (Blood and lymphatic system disorders) | 5
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 1
Pain: Abdomen NOS (Gastrointestinal disorders) | 1
Pain: Back (Musculoskeletal and connective tissue disorders) | 6
Pain: Bone (Musculoskeletal and connective tissue disorders) | 2
Pain: Breast (Reproductive system and breast disorders) | 1
Pain: Chest wall (Musculoskeletal and connective tissue disorders) | 1
Pain: Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain: Joint (Musculoskeletal and connective tissue disorders) | 2
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 3
Pain: Pain NOS (General disorders) | 3
Pain: Stomach (Gastrointestinal disorders) | 1
Pain: Testicle (Reproductive system and breast disorders) | 1
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 3
Platelets (Investigations) | 6
Sweating (diaphoresis) (General disorders) | 1
Vessel injury-vein: Other NOS (Vascular disorders) | 1
Vision-blurred vision (Eye disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Weight loss (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes